CLINICAL TRIAL: NCT07021209
Title: A Single-arm, Open-label, Phase I Clinical Study of GT719 Injection for Recurrent/Refractory Antibody-mediated Neurological Immune Diseases
Brief Title: GT719 Injection for Recurrent/Refractory Antibody-mediated Neurological Immune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-719-002
Record Dates: First submitted 2025-05-29; First posted 2025-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Neurological Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT719 Injection treatment group (Experimental): GT719 Injection
  Interventions: Biological: GT719 Injection

INTERVENTIONS:
Biological: GT719 Injection — GT719 Injection

SUMMARY:
This study is an open-label, prospective, exploratory clinical trial that includes a dose escalation phase and a dose expansion phase, aimed at evaluating the safety, cell dynamics, and preliminary efficacy of GT719 cells in adult participants with recurrent/refractory antibody-mediated neurological immune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily enrolled in the study, signed an informed consent form, willing and able to comply with the study protocol.
* Expected survival period>12 weeks.
* Any previous systemic treatment must have undergone at least 4 weeks or 5 half lives (whichever is shorter) by the time the participant plans to receive the study treatment.

Exclusion Criteria:

* History of organ transplantation, splenectomy, and allogeneic or autologous stem cell transplantation.
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to enrollment, requiring systemic anticoagulant therapy.
* Received systemic corticosteroids at a dose of ≥10 mg/day prednisone equivalent within 7 days prior to GT719 infusion, except for inhaled corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adversed events | 24 months
  To characterize the safety profile of GT719 in patients with recurrent/refractory antibody-mediated neurological immune diseases as measured by the incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics of GT719 cells | 24 months
  Survival time of GT719 cells after infusion of GT719 Injection

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Principal Investigator — Tongji Hospital; Daishi Tian, Principal Investigator — Tongji Hospital; Chuan Qin, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No